CLINICAL TRIAL: NCT02714907
Title: Clinical Data Validation of Novel Wireless Cortrium C3 Monitor for Continuous Electrocardiogram Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cortrium (Industry)
Collaborators: University Hospital Bispebjerg and Frederiksberg (Other); Aleris-Hamlet Hospitaler København (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: H-15006113
Record Dates: First submitted 2016-03-11; First posted 2016-03-22 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AF assessed from Cortrium C3 data (Experimental): Atrial fibrillation assessed from Cortrium C3 device data
  Interventions: Device: Cortrium C3 device; Device: Holter device
- AF assessed from Holter data (Experimental): Atrial fibrillation assessed from Holter data
  Interventions: Device: Cortrium C3 device; Device: Holter device

INTERVENTIONS:
Device: Cortrium C3 device — Data is read from Cortrium C3 monitor
Device: Holter device — Date is read from Holter device

SUMMARY:
The purpose of this study is to validate the quality of the ECG-signal acquired with the Cortrium C3 monitor. The intention is to evaluate whether the diagnosis of atrial fibrillation based on the ECG signal from the C3 monitor concurs with the current monitoring methods used in clinical practice.

DETAILED DESCRIPTION:
Development of new cost effective mobile devices and wireless technology has great potential in supervision of critically ill patients in wards as well as ambulant. Through continuous wireless monitoring in both the hospital and the patients home, detection of heart arrhythmias such as atrial fibrillation (AF) will be possible.

AF is the cause of a sizeable amount of strokes (15% of all, and more than 35% of the population over 80 years of age), which can be prevented through anticoagulation treatment if provided in time. Thus, many patients are referred to cardiologic ambulatory to be examined for AF, and are subjected to heart monitoring with a so-called Holter or event monitor. This entails the patient be equipped with several electrodes on the chest, to which leads are attached and connected to a sizable and bulky box. The patient carries this box around hanging from the shoulder, belt or something similar for one or several days. It is then required of the patient to come back and deliver the device, after which the data must be read and analysed, in order to work out a further plan for the patient. During admission, a similar system can be attached for continuous heart monitoring.

Cortrium (http://cortrium.com) has developed a wireless technology, where a small C3 monitor is attached to the chest with standard electrodes and the leads are built into the actual monitor. The quality of the signal has been tested on healthy adults, but is yet to be tested on patients suffering from arrhythmias

The purpose of this study is to validate the quality of the ECG-signal acquired with the Cortrium C3 monitor. The intention is to evaluate whether the diagnosis of atrial fibrillation based on the ECG signal from the C3 monitor concurs with the current monitoring methods used in clinical practice.

The measurements are performed on patients under investigation for AF at cardiology ambulatory Y at Frederiksberg-Bispebjerg Hospital and Aleris-Hamlet Hospital, Copenhagen. The patients are outfitted with a C3 monitor simultaneous with the use of the conventional ambulatory apparatus. This is a "Holter monitor" (Rozinn station RZ152+12 and RZ153+ from ScottCare Holter for Windows 2010 (CE0120) and "EventCare SA version" (CE0120), both bought via SEMCA Ap, Skævinge, Denmark.

Recordings with the usual apparatus are analysed in the usual fashion in the cardiology ambulatory. A copy of the recordings is registered anonymously and paired with the simultaneous recordings from the C3. The diagnosis is made by two observers, blinded to both patient identity and data source. Thus, data will not be personally identifiable. Validation is performed in collaboration with the department of cardiology.

Statistics:

With simultaneous supervision of 77 patients with increased incidence of AF it will be possible to determine whether the C3 is capable of detecting AF in at least 95% of the cases which Holter detects. Since the incidence of AF Is lower in the total patient group referred to Holter monitoring, we plan to include 150 patients to acquire the usable number of examinations.

Economic Conditions Helen Dominguez is the unfunded, and the responsible consultant of the study. Opeon Aps delivers C3 monitors for this clinical trial as well as brochure guides for patients and health care personnel. There are no economic benefits connected with the present clinical trial.

Publication of Results:

Opeon ApS (owner of Cortrium) is responsible for processing the material for publication of results in an international peer-reviewed journal as well as in the Danish popular scientific press related to new Medical equipment. Positive, negative and inconclusive results will be published.

Recruitment of Participants:

Patients who have planned ambulatory arrhythmia recording for diagnosis of intermittent AF will be asked by telephone to consider participating in the study.

After reading the participant information flyer, the subjects are invited to in-depth verbal information in the ambulatory. If the subjects accept to participate and provide a signed informed consent, they outfitted with a C3 monitor along with the standard Holter apparatus.

The study only includes subjects scheduled for Holter monitoring referred for atrial fibrillation examination, quantification of paroxysms, or heart rate during paroxysms.

Ethical Considerations:

Ethical Considerations: If the patient agrees to take part in the study, the main disadvantages are that it entails attachment of another three electrodes for the C3 monitor, increasing the risk of skin irritation, and receiving additional instructions for two devices. Since ECG recordings are non-invasive, and the C3 recordings do not result in further ambulatory visits than otherwise planned, we estimated that the strain on the patients is very limited.

The use of C3 for estimation of AF in future patients will decrease the trouble of loose leads. For this reason, using the C3 will also simplify the work of the healthcare personnel during the attachment procedure. Overall it may lead to an increase in quality as well as increase the capacity for examining cardiac arrhythmia in the cardiology ambulatory.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of atrial fibrillation
* Investigation of atrial fibrillation

Exclusion Criteria:

* Language difficulties
* Impaired cognitive function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2016-02; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation | Through study completion, an average of 3 months
  Expert readings of long-term ECG reports to assess number of AF paroxysms.
Heart rate (BPM) during atrial fibrillation | Through study completion, an average of 3 months
  Expert readings of long-term ECG reports to assess heart rate in BPM.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Helena, MD, PhD, Principal Investigator — Bispebjerg-Frederiksberg Hospitals
Locations (2):
- Denmark (2):
  - Department of Cardiology, Bispebjerg-Frederiksberg Hospitals, Frederiksberg
  - Aleris-Hamlet Private Hospital, Søborg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Saito T, Tamura K, Uchida D, Saito T, Togashi M, Nitta T, Sugisaki Y. Histopathological features of the resected left atrial appendage as predictors of recurrence after surgery for atrial fibrillation in valvular heart disease. Circ J. 2007 Jan;71(1):70-8. doi: 10.1253/circj.71.70. PMID 17186981
- [Background] Syed TM, Halperin JL. Left atrial appendage closure for stroke prevention in atrial fibrillation: state of the art and current challenges. Nat Clin Pract Cardiovasc Med. 2007 Aug;4(8):428-35. doi: 10.1038/ncpcardio0933. PMID 17653115
- [Background] Saltman AE, Gillinov AM. Surgical approaches for atrial fibrillation. Cardiol Clin. 2009 Feb;27(1):179-88, x. doi: 10.1016/j.ccl.2008.09.012. PMID 19111773
- [Background] Gillinov AM. Advances in surgical treatment of atrial fibrillation. Stroke. 2007 Feb;38(2 Suppl):618-23. doi: 10.1161/01.STR.0000247934.04848.79. PMID 17261702
- [Background] Al-Saady NM, Obel OA, Camm AJ. Left atrial appendage: structure, function, and role in thromboembolism. Heart. 1999 Nov;82(5):547-54. doi: 10.1136/hrt.82.5.547. PMID 10525506
- [Background] Fitzmaurice D. Atrial fibrillation and coagulation: who and when? Blood Rev. 2009 Nov;23(6):241-4. doi: 10.1016/j.blre.2009.07.006. Epub 2009 Aug 25. PMID 19709791
- [Background] Furberg CD, Psaty BM, Manolio TA, Gardin JM, Smith VE, Rautaharju PM. Prevalence of atrial fibrillation in elderly subjects (the Cardiovascular Health Study). Am J Cardiol. 1994 Aug 1;74(3):236-41. doi: 10.1016/0002-9149(94)90363-8. PMID 8037127
- [Background] Page RL, Wilkinson WE, Clair WK, McCarthy EA, Pritchett EL. Asymptomatic arrhythmias in patients with symptomatic paroxysmal atrial fibrillation and paroxysmal supraventricular tachycardia. Circulation. 1994 Jan;89(1):224-7. doi: 10.1161/01.cir.89.1.224. PMID 8281651
- [Background] Healey JS, Connolly SJ, Gold MR, Israel CW, Van Gelder IC, Capucci A, Lau CP, Fain E, Yang S, Bailleul C, Morillo CA, Carlson M, Themeles E, Kaufman ES, Hohnloser SH; ASSERT Investigators. Subclinical atrial fibrillation and the risk of stroke. N Engl J Med. 2012 Jan 12;366(2):120-9. doi: 10.1056/NEJMoa1105575. PMID 22236222
- [Background] Israel CW, Gronefeld G, Ehrlich JR, Li YG, Hohnloser SH. Long-term risk of recurrent atrial fibrillation as documented by an implantable monitoring device: implications for optimal patient care. J Am Coll Cardiol. 2004 Jan 7;43(1):47-52. doi: 10.1016/j.jacc.2003.08.027. PMID 14715182
- [Background] Thakkar S, Bagarhatta R. Detection of paroxysmal atrial fibrillation or flutter in patients with acute ischemic stroke or transient ischemic attack by Holter monitoring. Indian Heart J. 2014 Mar-Apr;66(2):188-92. doi: 10.1016/j.ihj.2014.02.009. Epub 2014 Mar 4. PMID 24814113
- [Background] Cotter PE, Martin PJ, Ring L, Warburton EA, Belham M, Pugh PJ. Incidence of atrial fibrillation detected by implantable loop recorders in unexplained stroke. Neurology. 2013 Apr 23;80(17):1546-50. doi: 10.1212/WNL.0b013e31828f1828. Epub 2013 Mar 27. PMID 23535493
- [Background] Sanna T, Diener HC, Passman RS, Di Lazzaro V, Bernstein RA, Morillo CA, Rymer MM, Thijs V, Rogers T, Beckers F, Lindborg K, Brachmann J; CRYSTAL AF Investigators. Cryptogenic stroke and underlying atrial fibrillation. N Engl J Med. 2014 Jun 26;370(26):2478-86. doi: 10.1056/NEJMoa1313600. PMID 24963567
- [Background] Fuster V, Ryden LE, Cannom DS, Crijns HJ, Curtis AB, Ellenbogen KA, Halperin JL, Le Heuzey JY, Kay GN, Lowe JE, Olsson SB, Prystowsky EN, Tamargo JL, Wann S; Task Force on Practice Guidelines, American College of Cardiology/American Heart Association; Committee for Practice Guidelines, European Society of Cardiology; European Heart Rhythm Association; Heart Rhythm Society. ACC/AHA/ESC 2006 guidelines for the management of patients with atrial fibrillation-executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the European Society of Cardiology Committee for Practice Guidelines (Writing Committee to Revise the 2001 Guidelines for the Management of Patients with Atrial Fibrillation). Eur Heart J. 2006 Aug;27(16):1979-2030. doi: 10.1093/eurheartj/ehl176. No abstract available. PMID 16885201
- [Background] Lazzaro MA, Krishnan K, Prabhakaran S. Detection of atrial fibrillation with concurrent holter monitoring and continuous cardiac telemetry following ischemic stroke and transient ischemic attack. J Stroke Cerebrovasc Dis. 2012 Feb;21(2):89-93. doi: 10.1016/j.jstrokecerebrovasdis.2010.05.006. Epub 2010 Jul 24. PMID 20656504
- [Background] Caldwell JC, Contractor H, Petkar S, Ali R, Clarke B, Garratt CJ, Neyses L, Mamas MA. Atrial fibrillation is under-recognized in chronic heart failure: insights from a heart failure cohort treated with cardiac resynchronization therapy. Europace. 2009 Oct;11(10):1295-300. doi: 10.1093/europace/eup201. Epub 2009 Aug 1. PMID 19648586
- [Background] Nyrnes A, Mathiesen EB, Njolstad I, Wilsgaard T, Lochen ML. Palpitations are predictive of future atrial fibrillation. An 11-year follow-up of 22,815 men and women: the Tromso Study. Eur J Prev Cardiol. 2013 Oct;20(5):729-36. doi: 10.1177/2047487312446562. Epub 2012 May 15. PMID 22588086
- [Background] Sulfi S, Balami D, Sekhri N, Suliman A, Kapur A, Archbold RA, Ranjadayalan K, Timmis AD. Limited clinical utility of Holter monitoring in patients with palpitations or altered consciousness: analysis of 8973 recordings in 7394 patients. Ann Noninvasive Electrocardiol. 2008 Jan;13(1):39-43. doi: 10.1111/j.1542-474X.2007.00199.x. PMID 18234005
- [Background] Paudel B, Paudel K. The diagnostic significance of the holter monitoring in the evaluation of palpitation. J Clin Diagn Res. 2013 Mar;7(3):480-3. doi: 10.7860/JCDR/2013/4923.2802. Epub 2013 Mar 1. PMID 23634400
- [Background] Hertzeanu H, Aron L. Holter monitoring for dizziness and syncope in old age. Acta Cardiol. 1985;40(3):291-9. PMID 3875198
- [Background] Hennersdorf MG, Schueller PO, Steiner S, Strauer BE. Prevalence of paroxysmal atrial fibrillation depending on the regression of left ventricular hypertrophy in arterial hypertension. Hypertens Res. 2007 Jun;30(6):535-40. doi: 10.1291/hypres.30.535. PMID 17664857
- Available data/document: Study Protocol — http://cortrium.com — In Danish language